CLINICAL TRIAL: NCT06647121
Title: A Randomized Pilot and Feasibility Trial Investigating a Mobile Application-Delivered Mindfulness Exercise for Navigating Psychological Distress: Dropping Anchor Delivered As a Stepwise Image Sequence
Brief Title: A Randomized Pilot Trial Investigating a Novel Mobile Application for Practicing Exercises from ACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbel Knauper (Other)
Responsible Party: Sponsor-Investigator, Barbel Knauper, James McGill Professor of Health Psychology, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB# 23-08-055
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Psychological Distress

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to condition assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT Workshop Plus ACTaide Mobile App (Experimental): In this condition, participants will attend a 1-hour virtual ACT psychoeducational workshop where they will learn about ACT, practice the dropping anchor exercise (with a guided image sequence), and learn how to use the ACTaide mobile app, which they will be asked to use to practice the dropping anchor exercise daily for two weeks. The main feature of the ACTaide app is the annotated image sequence to guide users through the steps of the exercise. The app also features customizable reminders notifications. Participants will receive three reminders per day encouraging them to practice the exercise.
  Interventions: Behavioral: ACT Psychoeducational Workshop; Behavioral: ACTaide Mobile App
- ACT Workshop Plus Reminders-only Mobile App (Active Comparator): In this condition, participants will attend a 1-hour virtual ACT psychoeducational workshop where they will learn about ACT, practice the dropping anchor exercise (without a guided image sequence), and learn how to use the reminders-only mobile app, which they will be asked to use to practice the dropping anchor exercise daily for two weeks. This app will not include the annotated image sequence from ACTaide and instead will only include customizable reminders notifications. Participants will receive three reminders per day encouraging them to practice the exercise.
  Interventions: Behavioral: ACT Psychoeducational Workshop; Behavioral: Reminders-only mobile app

INTERVENTIONS:
Behavioral: ACT Psychoeducational Workshop — The 1-hour ACT psychoeducational workshop will introduce participants to Acceptance and Commitment Therapy and include guided practice of the mindfulness exercise that they will be asked to practice for two weeks.
Behavioral: ACTaide Mobile App — The ACTaide mobile app is a novel app that is designed to support home practice of exercises from ACT via annotated image sequences and reminder notifications. A prototype version that features the dropping anchor mindfulness exercise will be investigated in this study.
  Arms: ACT Workshop Plus ACTaide Mobile App
Behavioral: Reminders-only mobile app — This app will include only reminder notifications to encourage home practice of the dropping anchor mindfulness exercise in the comparator condition. It will not include the annotated image sequence for the exercise (i.e., the primary feature of the ACTaide app to be investigated in the intervention condition).
  Arms: ACT Workshop Plus Reminders-only Mobile App

SUMMARY:
Mindfulness-related skills are associated with positive mental health outcomes and can be effectively taught through mobile apps. However, further research is needed to determine how best to support skill acquisition through the delivery of mindfulness exercises via smartphone apps. ACTaide is a novel mobile app designed to support home practice of mindfulness-related skills through exercises presented as stepwise annotated image sequences. The primary objective of this pilot and feasibility trial is to evaluate the feasibility of a prototype version of ACTaide. This two-arm parallel single-blinded (blinded participants) pilot trial will be conducted virtually with distressed Canadian adults. Participants (N = 60) will be recruited through the online platform Prolific. The intervention group will receive an Acceptance and Commitment Therapy (ACT) psychoeducational workshop and access to ACTaide for two weeks to support home practice of a mindfulness exercise from ACT: dropping anchor. The control group will receive the same psychoeducational workshop and access to a reminders-only mobile app to support their practice of the dropping anchor exercise. The main outcome measures will assess intervention feasibility, including adherence to the intervention, acceptability of the app, and retention rates. In addition, measures related to mindfulness-related skills and psychological distress will be collected. Prespecified progression criteria will be used to determine whether and how to proceed to a future trial designed to investigate the efficacy of ACTaide.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years old;
2. be fluent in English;
3. own a smartphone with a data plan;
4. report at least moderate psychological distress as measured by the 21-item Depression Anxiety Stress Scales (DASS-21; i.e., overall score of at least 43); and
5. report at least moderate motivation to learn a new psychotherapeutic exercise for navigating psychological distress (i.e., at least 6 out of 10).

Exclusion Criteria:

Due to the limited psychotherapeutic scope of the intervention, individuals were ineligible if they self-reported extremely severe psychological distress (i.e., an overall score of 82 or higher on the DASS-21) or a diagnosis of a severe mental illness (i.e., bipolar disorder, psychosis, schizophrenia, borderline personality disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Intervention adherence (home practice of mindfulness exercise) | 2 weeks
  the frequency and duration of home practice of a mindfulness exercise measured via the mobile app
ACTaide mobile app acceptability | 2 weeks
  an adapted version of the mHealth App Usability Questionnaire (MAUQ; Zhou et al., 2019) will be used to measure the acceptability of the app.
Participant retention | 4 weeks
  retention rates will be measured at the post-intervention and 2-week follow-up time points

SECONDARY OUTCOMES:
Changes in Symptoms of Depression, Anxiety, Stress | Changes in psychological distress will be measured from baseline to the 2-week, post-intervention time point, and from baseline to the four-week, follow-up time point.
  The 21-item Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995) will be included. It is the proposed primary outcome of future efficacy trials. The DASS-21 is a self-report measure that assesses individuals' symptoms of depression, anxiety, and stress in the past week. Participants are asked to indicate the extent to which each statement applied to them over the past week from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). Sample items include: "I found it hard to wind down" and "I felt down-hearted and blue." Scores for each subscale will be computed by taking the sum of all items from each respective subscale and multiplying by two. To assess the efficacy potential of the intervention, we calculate the proportion of participants in each condition that reported clinically meaningful reductions in psychological distress at the post-intervention and follow-up time points.
Changes in Mindfulness Skills | Changes in mindfulness skills will be measured from baseline to the two-week, post-intervention time point, and from baseline to the four-week, follow-up time point.
  Changes in mindfulness skills, a proposed secondary outcome for future efficacy trials, will be measured with the Multidimensional Psychological Flexibility Inventory Short Form (MPFI-24; Grégoire et al., 2020; Rolffs et al., 2018), which is a 24-item self-report questionnaire that assesses components of Psychological Flexibility and Inflexibility as defined by the Hexaflex model of ACT. The measure includes pairs of items that assess each of the six components of Psychological Flexibility (e.g., Acceptance, Present Moment Awareness) and Psychological Inflexibility (e.g., Experiential Avoidance, Lack of Contact with the Present Moment). In addition, two measures of equanimity will be included as potential secondary outcome measures for future efficacy trials: (1) the Even-mindedness subscale from the Two-Factor Equanimity Scale (Juneau et al., 2020), and the Equanimity Scale-16 (ES-16; Rogers et al., 2021).
Changes in Distress Tolerance | Changes in distress tolerance will be measured from baseline to the two-week, post-intervention time point and from baseline to the four-week, follow-up time point.
  The Distress Tolerance Scale short-form (DTS-SF; Gardner et al., 2018) will be included. It is a 4-item scale that measures individuals' perceived ability to experience, endure, and regulate negative psychological states. Participants in the present study will be asked to respond to each item based on their experiences over the past week; therefore, items were modified to past tense (example item: "I couldn't handle feeling distressed or upset.")

CONTACTS AND LOCATIONS:
Overall Officials: Bärbel Knäuper, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be uploaded to OSF after the completion of the study.
Supporting Information: Analytic Code
Time Frame: Data will be shared within approximately one year of the completion of data collection.
Access Criteria: Data will be available to all researchers via the OSF website.

REFERENCES:
- [Background] Di Sante J, Frayn M, Angelescu A, Knauper B. Proof-of-concept testing of a brief virtual ACT workshop for emotional eating. Appetite. 2024 Aug 1;199:107386. doi: 10.1016/j.appet.2024.107386. Epub 2024 Apr 30. PMID 38692511
- [Background] Dochat C, Wooldridge JS, Herbert MS, Lee MW, Afari N. Single-Session Acceptance and Commitment Therapy (ACT) Interventions for Patients with Chronic Health Conditions: A Systematic Review and Meta-Analysis. J Contextual Behav Sci. 2021 Apr;20:52-69. doi: 10.1016/j.jcbs.2021.03.003. Epub 2021 Mar 6. PMID 33868913
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Frayn M, Khanyari S, Knauper B. A 1-day acceptance and commitment therapy workshop leads to reductions in emotional eating in adults. Eat Weight Disord. 2020 Oct;25(5):1399-1411. doi: 10.1007/s40519-019-00778-6. Epub 2019 Sep 20. PMID 31541426
- [Background] Kazdin AE. Annual Research Review: Expanding mental health services through novel models of intervention delivery. J Child Psychol Psychiatry. 2019 Apr;60(4):455-472. doi: 10.1111/jcpp.12937. Epub 2018 Jun 13. PMID 29900543
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Background] Lewis M, Bromley K, Sutton CJ, McCray G, Myers HL, Lancaster GA. Determining sample size for progression criteria for pragmatic pilot RCTs: the hypothesis test strikes back! Pilot Feasibility Stud. 2021 Feb 3;7(1):40. doi: 10.1186/s40814-021-00770-x. PMID 33536076
- [Background] Linardon J, Fuller-Tyszkiewicz M. Attrition and adherence in smartphone-delivered interventions for mental health problems: A systematic and meta-analytic review. J Consult Clin Psychol. 2020 Jan;88(1):1-13. doi: 10.1037/ccp0000459. Epub 2019 Nov 7. PMID 31697093
- [Background] Linardon J, Torous J, Firth J, Cuijpers P, Messer M, Fuller-Tyszkiewicz M. Current evidence on the efficacy of mental health smartphone apps for symptoms of depression and anxiety. A meta-analysis of 176 randomized controlled trials. World Psychiatry. 2024 Feb;23(1):139-149. doi: 10.1002/wps.21183. PMID 38214614
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Patel V, Maj M, Flisher AJ, De Silva MJ, Koschorke M, Prince M; WPA Zonal and Member Society Representatives. Reducing the treatment gap for mental disorders: a WPA survey. World Psychiatry. 2010 Oct;9(3):169-76. doi: 10.1002/j.2051-5545.2010.tb00305.x. PMID 20975864
- [Background] Ronk FR, Korman JR, Hooke GR, Page AC. Assessing clinical significance of treatment outcomes using the DASS-21. Psychol Assess. 2013 Dec;25(4):1103-10. doi: 10.1037/a0033100. Epub 2013 Jun 3. PMID 23730826
- [Background] Zhou L, Bao J, Setiawan IMA, Saptono A, Parmanto B. The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study. JMIR Mhealth Uhealth. 2019 Apr 11;7(4):e11500. doi: 10.2196/11500. PMID 30973342